CLINICAL TRIAL: NCT06925035
Title: Efficacy of Combined 1927nm Thulium Fiber Laser and Supramolecular Salicylic Acid in Photoaging Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Weihui Zeng, Professor, Second Affiliated Hospital of Xi'an Jiaotong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023019
Record Dates: First submitted 2025-03-27; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-03

CONDITIONS: Photo-aged Skin; Laser
Keywords: Photoaging; supramolecular salicylic acid; Thulium Fiber Laser

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TFL-only group (Placebo Comparator): TFL Alone Treatment Side (Control/Placebo Side) Interventions:
  Pre-TFL Preparation:
  Topical application of Compound Lidocaine Cream (30-40 minutes) for anesthesia.Facial sterilization with alcohol.
  TFL Treatment:
  Half-face treatment with a 1927 nm fractional thulium fiber laser (WONTECH, Lavieen, South Korea).
  Parameters: Pulse energy 8-10 mJ, output power 10 W, pulse spacing 0.8 mm. Post-TFL Intervention:Immediate application of placebo (base material of 30% SSA) on the assigned facial side after TFL.Placebo gently massaged with saline for penetration simulation.
  Placebo maintained until clinical endpoint (mild erythema/whitening), followed by saline rinse and a 20-minute medical repair mask.
  Adjunctive Regimen (16 Weeks):
  Placebo applied biweekly (matching 30% SSA frequency) and daily (matching 2% SSA regimen).
  Interventions: Device: 1927nm fractional thulium fiber laser(TFL)
- PFL-SSA combination treatment group (Experimental): TFL-SSA Combination Therapy Side (Intervention Side) Interventions:
  Pre-TFL Preparation:
  Identical to the control side: Lidocaine Cream and alcohol sterilization.
  TFL Treatment:
  Same laser parameters and half-face coverage as the control side.
  Post-TFL Intervention:
  Immediate application of 30% SSA on the assigned facial side after TFL. SSA gently massaged with saline to enhance penetration. SSA maintained until clinical endpoint (erythema/whitening), followed by saline rinse and a 20-minute medical repair mask.
  Adjunctive Regimen (16 Weeks):
  30% SSA applied biweekly and 2% SSA applied daily to the combination therapy side.
  Interventions: Device: 1927nm fractional thulium fiber laser(TFL); Drug: supramolecular salicylic acid(SSA)

INTERVENTIONS:
Device: 1927nm fractional thulium fiber laser(TFL) — Prior to each session, Compound Lidocaine Cream (Beijing Ziguang Medication Manufacture Corporation Ltd.) was administered topically to the participants' faces for a duration of 30-40 minutes. Following sterilization with alcohol, the entire facial area was treated with a 1927 nm fractional thulium fiber laser (TFL) (WONTECH, Lavieen, South Korea). TFL parameters included a pulse energy of 8-10 mJ, an output power of 10 W, and a pulse spacing of 0.8 mm, ensuring comprehensive coverage of photodamaged regions.
Drug: supramolecular salicylic acid(SSA) — 30% SSA (SSA and placebo are provided by Broda ,Shanghai Rui Zhi Medicine Technology, Shanghai, China.) or placebo(the base material of 30% SSA) were randomly assigned to be applied on one side of the face immediately after completion of the 1927nm TFL treatment. The 30% SSA was maintained on facial skin until reaching the clinical endpoint, manifested as mild erythema and/or a characteristic frost-like epidermal whitening. Additionally, the combination therapy side of the subjects was treated with one session of 30% SSA biweekly and 2% SSA daily over a period of 16 weeks.
  Arms: PFL-SSA combination treatment group

SUMMARY:
Purpose: 1927nm fractional thulium fiber laser (TFL) has been shown to be effective in improving skin appearance by reducing pigmentation and loss of elasticity caused by photoaging. Supramolecular salicylic acid (SSA) has been utilized for chemical peeling with rejuvenation effect. This study aims to evaluate the effectiveness and safety of combined TFL and SSA treatment for photoaging.

Methods: Thirty-six patients with moderate-to-severe photoaging were enrolled and the two sides of the participants' face were randomly assigned to receive 30% SSA combined with TFL or TFL monotherapy. TFL was administered to both sides of the face on four occasions at four-week intervals, while the side receiving combined treatment additionally underwent eight chemical peels of 30% SSA fortnightly, supplemented by daily applications of 2% SSA. For the TFL-alone side, an equivalent dose of a placebo preparation was applied. The photographs, photoaging scores, melanin index (MI), erythema index (EI), skin hydration, trans-epidermal water loss (TEWL), dermal thickness, elasticity index, and skin rebound time were assessed.

DETAILED DESCRIPTION:
This prospective, split-face, randomized, double-blind clinical trial evaluated the efficacy of fractional thulium fiber laser (TFL) monotherapy versus TFL combined with topical succinic acid (SSA) for photoaging treatment. Eligible participants (aged 40-70 years) with symmetric facial photodamage and a modified photoaging scale score >11 were enrolled, excluding individuals with systemic diseases, skin pathologies, recent aesthetic treatments, or SSA allergies. Following ethical approval (MR-61-23-03452; 2023019) and informed consent, subjects underwent four TFL sessions (1927 nm, 8-10 mJ, 10 W, 0.8 mm spacing) at 4-week intervals. Post-TFL, one randomized facial side received 30% SSA (or placebo, biweekly) and 2% SSA (or vehicle, daily) for 16 weeks, with allocation blinded to participants and investigators. Interventions were standardized using a clinical endpoint of mild erythema/epidermal whitening, followed by saline rinsing and medical mask application. Preprocedural anesthesia with compound lidocaine cream and postoperative protocols (ice packs for adverse events, medical masks, sun protection, and delayed cleansing until scab detachment) were implemented. Adverse events and adherence to post-treatment care were monitored. The study adhered to Declaration of Helsinki principles, with anonymized data analysis and oversight by the ethics committee of the Second Affiliated Hospital of Xi'an Jiao Tong University.

ELIGIBILITY:
Inclusion Criteria:

- Enrolled patients were scored using the Modified Photodamage Scale (total score of 16), and subjects with a score greater than 11 were ultimately included (less than 4, mild; up to 4-8, moderate; up to 8-12, advanced; and greater than 12, severe photodamage).

Exclusion Criteria

* Severe systemic disease
* Skin tumours or infections
* Currently pregnant or breastfeeding
* Recent use (within the last 6 months) of oral or topical medications or phototherapy, laser, filler or botulinum toxin treatment
* Allergy to SA
* A history of keloid scarring.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
photodamage score | From enrollment to the end of treatment at 16 weeks
  Efficacy of photoaging improvement was assessed by the formula: ((Baseline photodamage score - Post-treatment photodamage score) / Baseline photodamage score) x 100%.All patients were photographed using a standardized digital camera (EOS 600D, Canon, Tokyo, Japan) under identical lighting conditions at each visit.Assessments were conducted at at weeks 0 (baseline), 4, 8, 12, and 16, ensuring consistent lighting and positioning. Photoaging scores were determined by three independent blinded dermatologists, utilizing a digital picture-contrast scale for grading. Distinct weighting factors were allocated to various photoaging characteristics.
  Photoaging scores were performed using a standardized scale named Photoaging Scale.And Photoaging score has a maximum value of 16 and a minimum value of 0.Lower photoaging scores mean more significant improvements after intervention.

SECONDARY OUTCOMES:
Melanin Index | Assessments were conducted at at weeks 0 (baseline), 4, 8, 12, and 16.
  utilizing the DermaLab® Combo (Cortex Technology).
Erythema Index | Assessments were conducted at at weeks 0 (baseline), 4, 8, 12, and 16.
  utilizing the DermaLab® Combo (Cortex Technology)
Transepidermal Water Loss | Assessments were conducted at at weeks 0 (baseline), 4, 8, 12, and 16.
  utilizing the DermaLab® Combo (Cortex Technology)
skin hydration | Assessments were conducted at at weeks 0 (baseline), 4, 8, 12, and 16.
  utilizing the DermaLab® Combo (Cortex Technology)
dermal thickness | Assessments were conducted at at weeks 0 (baseline), 4, 8, 12, and 16.
  utilizing the DermaLab® Combo (Cortex Technology)
elasticity index | Assessments were conducted at at weeks 0 (baseline), 4, 8, 12, and 16.
  utilizing the DermaLab® Combo (Cortex Technology)

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Xi'an Jiao Tong University, Xian, Shanxi, China